CLINICAL TRIAL: NCT03490266
Title: Robotic Versus Laparoscopic Ventral Hernia Repair: A Multicenter Randomized Controlled Trial
Brief Title: Robotic Versus Laparoscopic Ventral Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Shinil Shah, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-18-0137
Record Dates: First submitted 2018-03-21; First posted 2018-04-06 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Hernia, Ventral
Keywords: Ventral Hernia; Hernia Repair
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Laparoscopic Repair (Active Comparator): The abdomen will be entered and insufflated utilizing a 5 mm optical port. Only 5 mm ports will be utilized laterally to take down all anterior abdominal wall adhesions. A mid-density polypropylene mesh with a one-sided adhesion barrier that provides at least 5 cm of overlap in all directions will be inserted through a 11 or 12 mm port placed through the defect. Excision of hernia sac and preperitoneal fat and defect closure will be performed per current practice. The mesh will be secured in four points with 0-PDS sutures and/or tacked with a double crown of tacks per our current practice.
  Interventions: Procedure: Laparoscopic Repair
- Robotic Repair (Experimental): Three lateral ports will be placed including a 12 port for the camera. Adhesions will be taken down from the anterior abdominal wall. Hernia sac and preperitoneal fat will be excised per current practice and defect will be closed using a running locking barbed suture. A mid-density polypropylene mesh with a one-sided adhesion barrier that provides at least 5 cm of overlap in all directions will be inserted through the 12 mm port. The mesh will be secured circumferentially with a running barbed suture.
  Interventions: Procedure: Robotic Repair

INTERVENTIONS:
Procedure: Robotic Repair — The surgeon will be utilizing a robotic system to repair the hernia.
  Other Names: da Vinci Si Surgical System; Endoscopic Instrument Control System, Model IS3000
  Arms: Robotic Repair
Procedure: Laparoscopic Repair — The surgeon will be repairing the hernia laparoscopically.
  Arms: Laparoscopic Repair

SUMMARY:
Ventral hernias are a common disease and one half of all individuals are born with or will acquire a ventral hernia in their lifetime. Repair of ventral hernias may be associated with significant morbidity, including surgical site infection, hernia recurrence and reoperation. Minimally invasive ventral hernia repair decreases rates of surgical site infection and hospital length of stay, without affecting recurrence, however the laparoscopic approach to ventral hernia repair accounts for only about 1/3 of all total hernia repairs performed in the US. Recent large database studies have suggested that robotic ventral hernia repair may be associated with decreased hospital length of stay. However, this study is affected by common biases of database studies and randomized controlled trials are needed to assess the true impact of robotics for ventral hernia repair.

DETAILED DESCRIPTION:
Ventral hernias are a common disease and one-half of all individuals are born with or will acquire a ventral hernia in their lifetime. Repair of ventral hernias are associated with substantial morbidity including surgical site infection, hernia recurrence, and reoperation. Randomized controlled trials and nationwide databases have shown that minimally invasive ventral hernia repair (i.e. laparoscopic ventral hernia repair) as opposed to open ventral hernia repair is associated with decreased rates of surgical site infection and hospital length of stay with no impact on long-term outcomes of hernia recurrence.

Recent large database studies have suggested that robotic ventral hernia repair may be associated with decreased hospital length of stay. However, this study is affected by common biases of database studies and randomized controlled trials are needed to assess the true impact of robotics for ventral hernia repair.

The growth of the robotic platform in surgery is growing exponentially. Despite this, the evidence supporting robotics remains limited. Studies demonstrating benefit such as improved outcomes or decreased hospital length of stay, are largely cohort studies subject to substantial bias. Among randomized controlled trials, none have demonstrated benefit with robotic surgery.

Recently, the America's Hernia Society (AHS) has endorsed robotic ventral hernia surgery. A series of studies published under the AHS Quality Collaborative (AHSQC) database have demonstrated improved outcomes with robotic ventral hernia repair when compared to open and laparoscopic surgery. However, the results of these studies remain hypothesis generating and randomized controlled trials are needed.

This study would represent among the first randomized controlled trials assessing the effect of robotic versus laparoscopic ventral hernia repair.

ELIGIBILITY:
Inclusion Criteria:

-All patients undergoing elective ventral hernia repair deemed appropriate for minimally invasive repair.

Exclusion Criteria:

* Patients unlikely to survive beyond 2 years based upon surgeon judgment (e.g. advanced cirrhosis or metastatic cancer)
* Patients unlikely to follow-up (e.g. lives out of state or no phone)
* Advanced COPD or CHF
* History of open abdomen or extensive lysis of adhesions for bowel obstruction
* Ascites due to cirrhosis or malignancy
* Active infection such as infected mesh
* Ventral hernia size greater than 12 cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2022-05-12 (Actual)

PRIMARY OUTCOMES:
Total number of days in the hospital | 90 days post-operative
  Total number of days spent in the hospital. This will be calculated by adding the hospital length of stay for initial surgery, length of stay for any additional readmission resulting from the surgery, and emergency room visits resulting from the surgery. This information will be collected up to 90 days after the surgery.

SECONDARY OUTCOMES:
Surgical Site Infection (SSI) | post-operative at 1 month, 90 days, 1 year, 2 years, and 3 years
  CDC definition
Surgical Site Occurrence (SSO) | post-operative at 1 month, 90 days, 1 year, 2 years, and 3 years
  Hematoma, seroma, dehiscence, necrosis, non-healing wound found on abdominal exam.
Hernia Reoccurence | post-operative at 1 month, 90 days, 1 year, 2 years, and 3 years
  A hernia that was repaired in the past but has returned
Patient centered outcomes | post-operative at 1 month, 90 days, 1 year, 2 years, and 3 years
  Collected using HerQLes
Patient centered outcomes | post-operative at 1 month, 90 days, 1 year, 2 years, and 3 years
  Collected using EQ5D
Cost from a healthcare perspective | post-operative at 1 month, 90 days, 1 year, 2 years, and 3 years
  Looking at differences in what is spent for robotic repair and laparoscopic repair of ventral hernias

CONTACTS AND LOCATIONS:
Overall Officials: Shinil Shah, DO, Principal Investigator — UTHealth-Memorial Hermann; Mike K Liang, MD, Principal Investigator — UTHealth-Lyndon B. Johnson (LBJ) Hospital
Locations (2):
- United States (2):
  - UT Health-Memorial Hermann, Houston, Texas
  - UTHealth-Lyndon B. Johnson (LBJ) Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cherla DV, Moses ML, Viso CP, Holihan JL, Flores-Gonzalez JR, Kao LS, Ko TC, Liang MK. Impact of Abdominal Wall Hernias and Repair on Patient Quality of Life. World J Surg. 2018 Jan;42(1):19-25. doi: 10.1007/s00268-017-4173-6. PMID 28828517
- [Background] Liang MK, Holihan JL, Itani K, Alawadi ZM, Gonzalez JR, Askenasy EP, Ballecer C, Chong HS, Goldblatt MI, Greenberg JA, Harvin JA, Keith JN, Martindale RG, Orenstein S, Richmond B, Roth JS, Szotek P, Towfigh S, Tsuda S, Vaziri K, Berger DH. Ventral Hernia Management: Expert Consensus Guided by Systematic Review. Ann Surg. 2017 Jan;265(1):80-89. doi: 10.1097/SLA.0000000000001701. PMID 28009730
- [Background] Holihan JL, Alawadi Z, Martindale RG, Roth JS, Wray CJ, Ko TC, Kao LS, Liang MK. Adverse Events after Ventral Hernia Repair: The Vicious Cycle of Complications. J Am Coll Surg. 2015 Aug;221(2):478-85. doi: 10.1016/j.jamcollsurg.2015.04.026. Epub 2015 May 9. PMID 26206646
- [Background] Holihan JL, Hannon C, Goodenough C, Flores-Gonzalez JR, Itani KM, Olavarria O, Mo J, Ko TC, Kao LS, Liang MK. Ventral Hernia Repair: A Meta-Analysis of Randomized Controlled Trials. Surg Infect (Larchmt). 2017 Aug/Sep;18(6):647-658. doi: 10.1089/sur.2017.029. Epub 2017 May 30. PMID 28557648
- [Background] Holihan JL, Alawadi ZM, Harris JW, Harvin J, Shah SK, Goodenough CJ, Kao LS, Liang MK, Roth JS, Walker PA, Ko TC. Ventral hernia: Patient selection, treatment, and management. Curr Probl Surg. 2016 Jul;53(7):307-54. doi: 10.1067/j.cpsurg.2016.06.003. Epub 2016 Jun 18. No abstract available. PMID 27569431
- [Background] Carbonell AM, Warren JA, Prabhu AS, Ballecer CD, Janczyk RJ, Herrera J, Huang LC, Phillips S, Rosen MJ, Poulose BK. Reducing Length of Stay Using a Robotic-assisted Approach for Retromuscular Ventral Hernia Repair: A Comparative Analysis From the Americas Hernia Society Quality Collaborative. Ann Surg. 2018 Feb;267(2):210-217. doi: 10.1097/SLA.0000000000002244. PMID 28350568
- [Background] Prabhu AS, Dickens EO, Copper CM, Mann JW, Yunis JP, Phillips S, Huang LC, Poulose BK, Rosen MJ. Laparoscopic vs Robotic Intraperitoneal Mesh Repair for Incisional Hernia: An Americas Hernia Society Quality Collaborative Analysis. J Am Coll Surg. 2017 Aug;225(2):285-293. doi: 10.1016/j.jamcollsurg.2017.04.011. Epub 2017 Apr 24. PMID 28450062
- [Background] Prete FP, Pezzolla A, Prete F, Testini M, Marzaioli R, Patriti A, Jimenez-Rodriguez RM, Gurrado A, Strippoli GFM. Robotic Versus Laparoscopic Minimally Invasive Surgery for Rectal Cancer: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Ann Surg. 2018 Jun;267(6):1034-1046. doi: 10.1097/SLA.0000000000002523. PMID 28984644
- [Background] Tasiopoulou VS, Svokos AA, Svokos KA, Zacharoulis D, Magouliotis DE. Robotic versus laparoscopic sleeve gastrectomy: a review of the current evidence. Minerva Chir. 2018 Feb;73(1):55-63. doi: 10.23736/S0026-4733.17.07583-6. Epub 2017 Dec 14. PMID 29243456
- [Background] Ilic D, Evans SM, Allan CA, Jung JH, Murphy D, Frydenberg M. Laparoscopic and robotic-assisted versus open radical prostatectomy for the treatment of localised prostate cancer. Cochrane Database Syst Rev. 2017 Sep 12;9(9):CD009625. doi: 10.1002/14651858.CD009625.pub2. PMID 28895658
- [Background] Coakley KM, Sims SM, Prasad T, Lincourt AE, Augenstein VA, Sing RF, Heniford BT, Colavita PD. A nationwide evaluation of robotic ventral hernia surgery. Am J Surg. 2017 Dec;214(6):1158-1163. doi: 10.1016/j.amjsurg.2017.08.022. Epub 2017 Sep 20. PMID 29017732
- [Background] Muysoms FE, Miserez M, Berrevoet F, Campanelli G, Champault GG, Chelala E, Dietz UA, Eker HH, El Nakadi I, Hauters P, Hidalgo Pascual M, Hoeferlin A, Klinge U, Montgomery A, Simmermacher RK, Simons MP, Smietanski M, Sommeling C, Tollens T, Vierendeels T, Kingsnorth A. Classification of primary and incisional abdominal wall hernias. Hernia. 2009 Aug;13(4):407-14. doi: 10.1007/s10029-009-0518-x. Epub 2009 Jun 3. PMID 19495920
- [Derived] Dhanani NH, Lyons NB, Olavarria OA, Bernardi K, Holihan JL, Shah SK, Wilson TD, Loor MM, Kao LS, Liang MK. Robotic Versus Laparoscopic Ventral Hernia Repair: Two-Year Results From a Prospective, Multicenter, Blinded Randomized Clinical Trial. Ann Surg. 2023 Aug 1;278(2):161-165. doi: 10.1097/SLA.0000000000005903. Epub 2023 May 19. PMID 37203558
- [Derived] Dhanani NH, Olavarria OA, Holihan JL, Shah SK, Wilson TD, Loor MM, Ko TC, Kao LS, Liang MK. Robotic Versus Laparoscopic Ventral Hernia Repair: One-year Results From a Prospective, Multicenter, Blinded Randomized Controlled Trial. Ann Surg. 2021 Jun 1;273(6):1076-1080. doi: 10.1097/SLA.0000000000004795. PMID 33630447
- [Derived] Olavarria OA, Bernardi K, Shah SK, Wilson TD, Wei S, Pedroza C, Avritscher EB, Loor MM, Ko TC, Kao LS, Liang MK. Robotic versus laparoscopic ventral hernia repair: multicenter, blinded randomized controlled trial. BMJ. 2020 Jul 14;370:m2457. doi: 10.1136/bmj.m2457. PMID 32665218